CLINICAL TRIAL: NCT05295134
Title: A Randomised, Double-Blind, Placebo Controlled, Dose Ranging Study to Investigate the Safety & Efficacy of Candida Rugosa Lipase on Reduction of Serum Triglyceride
Brief Title: Effect of Candida Rugosa Lipase on Serum Triglyceride Lowering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BIO-CAT, Inc. (Industry)
Collaborators: Atlantia Food Clinical Trials (Industry); Cork University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AFCRO-047
Record Dates: First submitted 2022-03-11; First posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Hypertriglyceridemia
Keywords: triglyceride; lipase; cholesterol; cylindracea; rugosa; digestion; triacylglycerol
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Lip4 protein, Candida rugosa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo
- Lipase: Low-Dose (Active Comparator): Candida cylindracea lipase (75,000 FIP per serving)
  Interventions: Dietary Supplement: Candida cylindracea lipase (225,000 FIP lipase units per day)
- Lipase: Medium-Dose (Active Comparator): Candida cylindracea lipase (150,000 FIP per serving)
  Interventions: Dietary Supplement: Candida cylindracea lipase (450,000 FIP lipase units per day)
- Lipase: High-Dose (Active Comparator): Candida cylindracea lipase (225,000 FIP per serving)
  Interventions: Dietary Supplement: Candida cylindracea lipase (675,000 FIP lipase units per day)

INTERVENTIONS:
Dietary Supplement: Placebo — Participants were directed to consume 1 placebo capsule containing maltodextrin, three times daily, for 90 days. Subjects were directed to consume the capsules with their three largest eating occasions of the day.
  Arms: Placebo
Dietary Supplement: Candida cylindracea lipase (225,000 FIP lipase units per day) — Participants were directed to consume 1 capsule containing lipase (75,000 FIP lipase units per capsule), three times daily, for 90 days. Subjects were directed to consume the capsules with their three largest eating occasions of the day.
  Other Names: GFA-918; Candida rugosa lipase
  Arms: Lipase: Low-Dose
Dietary Supplement: Candida cylindracea lipase (450,000 FIP lipase units per day) — Participants were directed to consume 2 capsules containing lipase (75,000 FIP lipase units per capsule), three times daily, for 90 days. Subjects were directed to consume the capsules with their three largest eating occasions of the day.
  Other Names: GFA-918; Candida rugosa lipase
  Arms: Lipase: Medium-Dose
Dietary Supplement: Candida cylindracea lipase (675,000 FIP lipase units per day) — Participants were directed to consume 2 capsules containing lipase (112,500 FIP lipase units per capsule), three times daily, for 90 days. Subjects were directed to consume the capsules with their three largest eating occasions of the day.
  Other Names: GFA-918; Candida rugosa lipase
  Arms: Lipase: High-Dose

SUMMARY:
The primary objective of this study was to evaluate the safety and tolerability of 3 doses of fungal lipase in the treatment of adults with mildly elevated serum triglycerides. The secondary objective was to assess the efficacy of fungal lipase in reducing serum triglycerides in adults with mildly elevated serum triglycerides.

DETAILED DESCRIPTION:
According to the World Health Organization, ischemic heart diseases and stroke were the leading causes of death globally in 2019, accounting for 16% and 11% of the world's total deaths, respectively. The American Heart Association reported in 2020 that approximately 87% of all strokes are ischemic strokes, in which blood flow to the brain is blocked (Virani et al). That blockage is typically caused by an accumulation of fatty deposits inside triglycerides (atherosclerosis). Higher levels of serum triglycerides are linked to an increased risk of ischemic stroke in men and women. Researchers tracked 7,579 women and 6,372 men whose triglyceride and cholesterol measurements were taken in the late 1970s. Subjects were followed for up to 33 years. During the follow-up period, 837 women and 837 men developed ischemic stroke. Both men and women had a higher risk of stroke with high levels of triglycerides, in particular triglyceride levels of 5 mmol/L (443 mg/dL or 5.0 mmol/L) or more. These individuals carried four-fold greater stroke risk than those with lower levels (Varbo et al).

Each of the current treatments for hypertriglyceridemia has negative side effects and therefore many individuals that suffer from this condition decline treatment to reduce stroke risk. Oral supplementation with a fungal lipase preparation from Candida cylindracea (formerly rugosa), commonly found in dietary supplements for digestive health, is a candidate strategy to lower triglycerides without side effects.

During digestion, each of lingual, gastric, and pancreatic lipases combine to remove the outer 2 fatty acids from ingested, dietary triglycerides, thus forming monoglycerides and 2 free fatty acids. Following uptake by intestinal enterocytes, the free fatty acids are re-esterified with the monoglycerides to reform triglycerides before release in to the bloodstream. Overconsumption of dietary fats can thus lead to elevated levels of serum triglycerides.

Candida cylindracea (formerly rugosa) lipase, however, hydrolyzes all three fatty acids from dietary triglycerides to release free fatty acids and the glycerol backbone. It is predicted that most of these free fatty acids and glycerol molecules enter the bloodstream without reformation to triglycerides by the major metabolic pathway to reform the triglycerides from monoglycerides. Nonetheless, an alternate metabolic pathway to generate triglycerides from free fatty acids alone does exist in enterocytes.

The investigators tested the hypothesis that fungal lipase-mediated lowering of dietary monoglycerides would lower serum triglyceride levels in a randomized, double-blind, placebo controlled parallel arm clinical trial of 39 subjects with elevated serum triglyceride levels. Subjects were between 18 and 75 years of age, with good general health and mildly elevated serum triglycerides (150 mg/dL to 500 mg/dL, or 1.7 mmol/L to 5.6 mmol/L). The study included 4 study site visits over a 13 to 16 week period (including baseline period).

Subjects underwent an initial phone screen and were asked questions regarding their age and general health. Eligible subjects were scheduled for a screening visit. Subjects attend all visits in a fasted state. At the screening visit (Visit 1), the inclusion and exclusion criteria were reviewed and the overall details of the study were explained and informed consent was obtained. Blood pressure, body weight, and body mass index (BMI) were measured. Family and medical history and general health were recorded.

A fasting blood sample was collected and serum triglycerides were measured. Subjects with serum triglyceride levels between 151 mg/dL (1.71 mmol/L) and 499 mg/dL (5.65 mmol/L) were invited to participate in the study. Eligible subjects were scheduled to return to the study site within 4 weeks for their baseline visit (Visit 2).

At Visit 2, a fasting blood sample (12 mL) was collected for glucose, electrolyte, triglyceride, cholesterol (including HDL, LDL, VLDL), liver and kidney function, and HbA1C measurements. Subjects were randomized to one of 4 arms: 1) placebo (n = 9), 2) 1X low-dose (n = 10), 3) 2X medium-dose (n = 10), and 4) 3X high-dose (n = 10). Subjects were provided with a 90 day supply of investigational study product (lipase or placebo) and were instructed to take one dose with each major meal (3 doses per day) for the next 90 days. Subjects were instructed to follow their standard diet and exercise routine for the duration of the study. Subjects were scheduled to return to the study site after 30 days (+/- 4 days) for Visit 3.

At Day 30 (Visit 3), a fasting blood sample (12 mL) was collected for glucose, electrolytes, triglyceride, cholesterol (including HDL, LDL, VLDL), liver and kidney function, and HbA1C measurements. Subjects were scheduled to return to the study site for the 4th and final visit at Day 90. At Day 90, a fasting blood sample (12 mL) was collected for glucose, electrolyte, triglyceride, cholesterol (including HDL, LDL, VLDL), liver and kidney function, and HbA1C measurements. Subjects returned any unused study product and compliance was assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent
2. Be between 18 and 75 years of age
3. Be in generally good health as determined by the investigator
4. Serum triglyceride levels between 151 mg/dL (1.71 mmol/L) and 499 mg/dL (5.65 mmol/L)

Exclusion Criteria:

1. Are less than 18 and greater than 75 years of age
2. Females are pregnant, lactating or wish to become pregnant during the study
3. Are hypersensitive to any of the components of the test product,
4. Have a significant acute or chronic, unstable and untreated disease or any condition which contraindicates, in the investigator's judgement, entry to the study
5. Have an active gastrointestinal disorder or previous gastrointestinal surgery
6. Have a known family history of hyperlipidemia
7. Having a condition or have taken a medication or supplement that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results, including triglyceride lowering medications (e.g., fibrates and statins) and supplements (e.g., plant sterols/stanols, fish oil supplements, and vitamin B complex supplements)
8. Have not made any major dietary changes in the past 3 months
9. History of illicit drug use
10. Subjects who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial
11. Subjects may not be receiving treatment involving experimental drugs
12. If the subject has participated in a recent experimental trial, the trial must have been completed not less than 60 days prior to this study
13. Have a malignant disease or any concomitant end-stage organ disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2014-10-06 (Actual); Study Completion 2014-11-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events | 90 days
  Self-reported adverse events at Visits 1, 2, and 3

SECONDARY OUTCOMES:
The change in levels of fasting serum triglycerides | 90 days
  Serum triglycerides (mmol/L)
The change in blood levels of fasting cholesterol | 90 days
  HDL cholesterol (mmol/L), LDL cholesterol (mmol/L), and total cholesterol (mmol/L)
Safety: Glycated hemoglobin A1C (HbA1C) | 90 days
  Blood HbA1C (mmol/mol)
Safety: Glucose | 90 days
  Blood glucose (mmol/L)
Safety: Alanine aminotransferase (ALT) | 90 days
  Blood ALT (IU/L)
Safety: Aspartate aminotransferase (AST) | 90 days
  Blood AST (IU/L)
Safety: Alkaline phosphatase (ALP) | 90 days
  Blood ALP (IU/L)
Safety: Gamma-glutamyl transferase (GGT) | 90 days
  Blood GGT (IU/L)
Safety: Sodium | 90 days
  Blood sodium (mEq/L)
Safety: Potassium | 90 days
  Blood potassium (mEq/L)
Safety: Chloride | 90 days
  Blood chloride (mmol/L)
Safety: Calcium | 90 days
  Blood calcium (mmol/L)
Safety: Phosphate | 90 days
  Blood phosphate (mmol/L)
Safety: Magnesium | 90 days
  Blood magnesium (mmol/L)
Safety: Urea | 90 days
  Blood urea (mmol/L)
Safety: Creatinine | 90 days
  Blood creatinine (umol/L)
Safety: Total protein | 90 days
  Blood total protein (g/L)
Safety: Albumin | 90 days
  Blood albumin (g/L)
Safety: Globulin | 90 days
  Blood globulin (g/L)
Safety: Total bilirubin | 90 days
  Blood total bilirubin (umol/L)
Safety: Uric acid | 90 days
  Blood uric acid (umol/L)
36-Item Short Form Health Survey (SF-36) | 90 days
  Physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH), physical component summary (PCS), mental component summary (MCS)

CONTACTS AND LOCATIONS:
Overall Officials: Fergus Shanahan, MD, PhD, Principal Investigator — Cork University Hospital
Locations (1):
- Atlantia Food Clinical Trials, Western Gateway Bldg, University College Cork, Cork, Co. Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Varbo A, Nordestgaard BG, Tybjaerg-Hansen A, Schnohr P, Jensen GB, Benn M. Nonfasting triglycerides, cholesterol, and ischemic stroke in the general population. Ann Neurol. 2011 Apr;69(4):628-34. doi: 10.1002/ana.22384. Epub 2011 Feb 18. PMID 21337605
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061